CLINICAL TRIAL: NCT03774316
Title: De-escalation of Antifungal Treatment in Immunocompromised Critically Ill Patients With Suspected Invasive Candida Infection: Incidence, Associated Factors, and Safety
Brief Title: De-escalation - Antifungal Treatment Immunocompromised Patients
Acronym: D-ATFIM
Status: Completed | Type: Observational
Sponsor: University Hospital, Lille (Other)
Responsible Party: Sponsor
Other Study IDs: 2017_32; 2017-A03113-50 (Other: ID-RCB number, ANSM)
Record Dates: First submitted 2018-12-03; First posted 2018-12-12 (Actual); Last update posted 2025-12-23 (Actual); Status verified 2025-12

CONDITIONS: Invasive Fungal Disease; Critical Illness
Keywords: De-escalation; Antifungal treatment; Mortality; Immunocompromised; Intensive care
MeSH Terms: conditions — Invasive Fungal Infections; Critical Illness

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
A small proportion of intensive care unit patients receiving antifungals have a proven invasive fungal infection. However, antifungal treatment has side effects such as toxicity, emergence of resistance, and high cost. Moreover, empirical antifungal treatment is still a matter for debate in these patients. Our study aimed to determine the incidence, associated factors, and safety of de-escalation of antifungals in immunocompromised critically ill patients.

This prospective observational study is conducted in 14 ICU, during a 6 months period. All immunocompromised patients hospitalized for >5d and treated with antifungals for suspected or proven invasive candida infection will be included De-escalation is defined as a reduction in antifungal spectrum or stopping initial drugs within the 5 days following their initiation. The three antifungals considered in this study are from the narrowest to the widest spectrum: fluconazole, caspofungin and liposomal amphotericin B.

DETAILED DESCRIPTION:
This is a retrospective and prospective observational multicenter study, aiming to determine the incidence, and safety of antifungal de-escalation in immunocompromised patients, and also factors associated with de-escalation.

ELIGIBILITY:
Inclusion Criteria:

* Adults immunocompromised patients hospitalized in intensive care units
* Predictable invasive mechanical ventilation duration > 96h
* Signed consent (by patient or its representative)
* First antifungal treatment initiation in ICU for proven or suspected candida infection

Exclusion Criteria:

* Pregnant or breast-feeding women.
* Fungal infection other than invasive candida
* Prophylactic antifungal treatment.
* Lack of informed consent
* Predictable mechanical ventilation duration less than 48 hours
* Patients discharged from ICU before the 5th day after initiation of TAF

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adults immunocompromised patients hospitalized in intensive care units (Age ≥18 years)
  Immunosuppression is defined by:
  * long-term immunosuppressive therapy (> 3 months) or high-dose corticosteroid therapy (> 0.5 mg / kg / day for at least 3 days)
  * Solid organ transplant
  * Solid cancer (active or in remission since <5 years)
  * Malignant haemopathy
  * HIV infection with CD4 <200
Sampling Method: Non-Probability Sample
Enrollment: 275 (Actual)
Dates: Start 2019-01-28 (Actual); Primary Completion 2023-11-07 (Actual); Study Completion 2023-11-07 (Actual)

PRIMARY OUTCOMES:
Percentage of patients with de-escalation of antifungal treatment | 5 days following start of antifungal treatment
  De-escalation is defined as a reduction in antifungal treatment spectrum (switch from echinocandines or Amphotericin B to Azoles) or stopping all antifungals within the 5 days following their initiation

SECONDARY OUTCOMES:
Risk factors for de-escalation of antifungal therapy | during the 5 days following start of antifungal
  Clinical characteristics and conditions significantly associated with de-escalation by univariate analysis will be entered in a multiple regression model to determine those independently associated with de-escalation
Number of days free of mechanical ventilation | until day 28 after start of antifungal treatment
  days with no mechanical ventilation
Number of days free of antifungal treatment | until day 28 after start of antifungal treatment
  days with no antifungal treatment
Length of ICU stay | until day 28 after start of antifungal treatment
  days in the ICU
All-cause mortality | until day 28 after start of antifungal treatment
  mortality related to any cause
Percentage of patients with reoccurrence of candidiasis | until day 7 after stop of antifungal treatment
  reccurrence of candidiasis is defined as a new episode after the end of antifungal treatment

CONTACTS AND LOCATIONS:
Overall Officials: Saad Nseir, MD,PhD, Principal Investigator — University Hospital, Lille
Locations (1):
- CHU Lille, Lille, France